CLINICAL TRIAL: NCT03608670
Title: Extravascular ICD Pilot Study
Acronym: EV ICD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDT17034
Record Dates: First submitted 2018-06-12; First posted 2018-08-01 (Actual); Results first posted 2022-04-22 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Tachycardia; Ventricular Arrythmia
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): Patients will be implanted with an extravascular ICD and undergo requisite electrical testing.
  Interventions: Device: Defibrillation using the Extravascular ICD

INTERVENTIONS:
Device: Defibrillation using the Extravascular ICD — VT/VF induction attempted for defibrillation testing, as well as requisite electrical testing.

SUMMARY:
The proposed study is designed to characterize the safety and efficacy of a new extravascular implantable cardioverter defibrillator (ICD) system in humans.

DETAILED DESCRIPTION:
The study will recruit male and female adult subjects that meet all of the inclusion criteria and none of the exclusion criteria. All subjects will be indicated to receive an ICD.

The EV ICD system will be implanted and the subjects will be followed for at least 3 months following implantation of the system.

Subjects will be exited after follow-up is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a Class I or IIa indication for implantation of an ICD according to the ACC/AHA/HRS Guidelines[1]
2. Patient is willing and able to sign and date the Informed Consent Form.
3. Patient is at least 18 years of age and meets age requirements per local law
4. Patient is geographically stable and willing and able to comply with the study procedures and visits for the duration of the follow-up

[1] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Hlatky MA, Granger CB, Hammill SC, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS guideline for management of patients with ventricular arrhythmias

-

Exclusion Criteria:

1. Patient has indications for bradycardia pacing [1] or Cardiac Resynchronization Therapy (CRT) [2] (Class I, IIa, or IIb indication)
2. Patient has an existing or had a prior pacemaker, ICD, or CRT device implant or leads
3. Patient has anatomical abnormality that significantly increases implant risk[3] including:

   • Severe obesity [4]
   * Marked RV dilation
   * Marked sternal abnormality
   * Hiatus hernia that distorts mediastinal anatomy
4. Patient has prior chest radiotherapy
5. Patient had previous mediastinitis
6. Patient had previous coronary artery bypass grafting procedure
7. Patient has existing transcatheter aortic valve replacement
8. Patient has gastrostomy tube
9. Patient has had a prior sternotomy, prior mediastinal instrumentation, prior abdominal surgery in the epigastric region, or planned sternotomy
10. Patient has previous pericarditis that:

    • Was chronic and recurrent, or

    • Resulted in pericardial effusion [5], or

    • Resulted in pericardial thickening or calcification [6]
11. Patients with a medical condition that precludes them from undergoing defibrillation testing, such as:

    • known LV thrombus

    • decompensated heart failure
    * LVEF <20% [7]
    * other physician discretion
12. Patient has persistent Atrial Fibrillation who is at high risk of a thromboembolic event with a CHA₂DS₂-VASc score ≥3, or is contraindicated for having anticoagulation interrupted for ≥72 hours
13. Patients with comorbidities which may increase surgical risk of complications[8] including:

    • severe aortic stenosis
    * COPD and is oxygen dependent
    * Hepatosplenomegaly
    * Marked hepatomegaly
14. Patient is on renal dialysis
15. Patient with any evidence of active infection or undergoing treatment for an infection
16. Patient with current implantation of neurostimulator or any other chronically implanted device which uses current in the body.
17. Patients with a limited life expectancy of less than 12 months
18. Patient is enrolled or planning to enroll in a concurrent drug or device study that may confound the results of this study, without documented pre-approval from a Medtronic study manager
19. Patient with any exclusion criteria as required by local law (e.g., age, pregnancy, breast feeding)
20. Pregnant women or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth regulation method or abstinence [9]

[1] 2015 HRS/EHRA/APHRS/SOLAECE expert consensus statement on optimal implantable cardioverter-defibrillator programming and testing).

[2] ACC/AHA/HRS guidelines for Cardiac Resynchronization Therapy [3] Per physician discretion [4] BMI > 40 [5] As documented on echo or MRI [6] As documented on CT scan or MRI [7] Most recent LVEF in the last 180 days (inclusive) [8] Per physician discretion [9] if required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to EV ICD Pilot Study procedures

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Crozier, MB ChB, Principal Investigator — Christchurch Hospital, Christchurch, New Zealand
Locations (4):
- Australia (3):
  - The Prince Charles Hospital, Brisbane
  - MonashHeart, Clayton
  - Austin Health, Heidelberg
- Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crozier I, Haqqani H, Kotschet E, Shaw D, Prabhu A, Roubos N, Alison J, Melton I, Denman R, Lin T, Almeida A, Portway B, Sawchuk R, Thompson A, Sherfesee L, Liang S, Lentz L, DeGroot P, Cheng A, O'Donnell D. First-in-Human Chronic Implant Experience of the Substernal Extravascular Implantable Cardioverter-Defibrillator. JACC Clin Electrophysiol. 2020 Nov;6(12):1525-1536. doi: 10.1016/j.jacep.2020.05.029. Epub 2020 Aug 26. PMID 33213813

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 26 participants consented and enrolled into the protocol. 5 participants were exited prior to an implant attempt.
Groups:
- Experimental: Patients enrolled to receive an extravascular ICD and undergo requisite electrical testing.
  Defibrillation using the Extravascular ICD: VT/VF induction attempted for defibrillation testing, as well as requisite electrical testing.
Period: Overall Study
Arm/Group | Experimental
Started | 26
Implant Attempted | 21
Successfully Implanted | 17
2-week Follow-up | 17
4-6 Weeks Follow-up | 17
Completed (Completed 3 Months follow-up for primary safety objective.) | 16
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White or Caucasian | 22
  Other: Maori | 2
  Other: Macedonian | 1
  Other: Afghani | 1
ICD Indication [Count of Participants; unit: Participants] — NYHA Functional Class grading:
  Class I: No limitations. Ordinary physical activity does not cause undue fatigue, dyspnoea or palpitations (asymptomatic LV dysfunction). Class II: Slight limitation of physical activity. Ordinary physical activity results in fatigue, palpitation, dyspnoea or angina pectoris (mild). Class III: Marked limitation of physical activity. Less than ordinary physical activity leads to symptoms (moderate). Class IV: Unable to carry on any physical activity without discomfort. Symptoms of CHF present at rest (severe).
  Participants
    Class I indication: Cardiac arrest due to VF/hemodynamically unstable sustained VT | 4
    Class I indication: Structural heart disease and spontaneous sustained VT | 1
    Class I indication: LVEF ≤ 35% due to prior MI, NYHA Class II or III | 5
    Class I indication: Nonischemic dilated cardiomyopathy, LVEF ≤ 35%, NYHA Class II or III | 5
    Class IIa indication: LV dysfunction due to prior MI, LVEF ≤ 30%, NYHA Class I | 3
    Class I Indication: Hypertrophic cardiomyopathy, 1 or more major risk factors for SCD | 6
    Class I Indication: Arrhythmogenic RV dysplasia / cardiomyopathy, ≥ 1 risk factor for SCD | 1
    Class IIb indication: Nonischemic heart disease, LVEF ≤ 35%, NYHA functional Class I | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Outcome - Number of Participants That Had Successful Termination of Ventricular Fibrillation Episodes at Implantation
Description: Each subject will demonstrate a successful defibrillation outcome if either 2 successive induced ventricular fibrillation episodes are terminated by the subject's device delivering a shock at the required energy level, or if one such episode is successfully terminated by the subject's device delivering a shock at a lower energy level. Up to 5 such episodes may be induced to test device efficacy.
Time Frame: At Implantation
Population: Number of participants who underwent and completed the defibrillation testing protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 20
Participants | 18

2. Primary Outcome: Safety Outcome - Percentage of Participants With Freedom From Major System and Procedure Related Complications at 3 Months (90 Days)
Description: Subjects will be monitored to determine whether they experience a major procedure- or system-related complication within 3 months (90 days) post-implant.
Time Frame: 3 months (90 days)
Population: All participants for whom an implant of the investigational product was attempted were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental
Number analyzed (Participants) | 21
percentage of participants | 94.1 [83.6 to 100]

ADVERSE EVENTS:
Time Frame: Assessed from Implant visit through to 3 Months (90 days inclusive)
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=21)
Lead dislodgement (Product Issues) | 2 (2) — Includes one lead dislodgement unrelated to the EV ICD
Orthostatic hypotension (Vascular disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=21)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Implant site swelling (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03608670/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03608670/SAP_001.pdf